CLINICAL TRIAL: NCT07105358
Title: Vision Improvement Through Behavioral Rehabilitation And Neuroplasticity Training
Brief Title: Visual Plasticity Following Brain Lesions
Acronym: VIBRANT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00008292
Record Dates: First submitted 2025-07-11; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Visual Field Defect; Stroke; Hemianopia; Quadrantanopia; Cortical Blindness; Brain Tumor; Traumatic Brain Injury; Visual Field Defect, Peripheral
MeSH Terms: conditions — Stroke; Hemianopsia; Blindness, Cortical; Brain Neoplasms; Brain Injuries, Traumatic | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: 1. Initial 2-Day Sessions: Participants receive either real or sham transcranial random noise stimulation (tRNS) combined with perceptual learning-based training.
  2. Washout Period: A minimum 1-week washout period (typically around 2 weeks) is included to minimize potential carry-over effects.
  3. Final 2-Day Sessions: Participants complete the alternate stimulation condition (sham or real) paired with perceptual learning-based training.
Who Masked: Participant, Investigator
Masking Description: This study is double-blind, meaning that both the participants and the researchers will be blinded to the treatment conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- tRNS with perceptual learning-based training (Experimental): Each 2-day session consists of up to three 18-minute transcranial random noise stimulation (tRNS) paired with perceptual learning-based training.
  Interventions: Device: transcranial random noise stimulation (tRNS); Behavioral: Perceptual learning-based training
- Sham with perceptual learning-based training (Sham Comparator): Each 2-day session consists of up to three 18-minute sham stimulation paired with perceptual learning-based training.
  Interventions: Device: Sham Stimulation; Behavioral: Perceptual learning-based training

INTERVENTIONS:
Device: transcranial random noise stimulation (tRNS) — Stimulation location: bilateral human middle temporal complex (hMT+). Stimulation parameters: 1 mA current intensity, with a frequency range of 101-640 Hz.
  Arms: tRNS with perceptual learning-based training
Device: Sham Stimulation — Stimulation location: bilateral human middle temporal complex (hMT+). Stimulation parameters: Ramp up stimulation at 1mA with a frequency range of 101-640Hz for the first 30 seconds followed by no current for the remainder of the duration.
  Arms: Sham with perceptual learning-based training
Behavioral: Perceptual learning-based training — A motion discrimination task, judging the global direction of moving dot stimuli with two different coherence levels.

SUMMARY:
The VIBRANT (Vision Improvement through Behavioral Rehabilitation And Neuroplasticity Training) study is a prospective, double-blind, crossover design (within-subject) in participants with homonymous hemianopia-a type of visual field loss resulting from damage to the post-chiasmatic visual pathways. It aims to investigate whether transcranial random noise stimulation (tRNS) combined with perceptual learning-based training has potential for improving visual impairments.

ELIGIBILITY:
A. Stroke, brain tumor, or traumatic brain injury patients

Inclusion Criteria:

1. At least 18 years of age.
2. Capable of providing informed consent and complying with study procedures.
3. Unilateral or bilateral focal brain damage causing loss of vision.
4. At least three months post-stroke or traumatic brain injury, or a stable brain tumor within the past year.

Exclusion Criteria:

1. Severe CNS diseases or disorders unrelated to the focal lesion, which could interfere with study results.
2. Severe mental health challenges that could interfere with study results, or current or recent (within the past 6 months) drug or alcohol abuse or addiction as defined by DSM-5.
3. Vision loss resulting from ocular disease or disorder.

B. Healthy volunteers (age-matched controls):

Inclusion Criteria:

1. At least 18 years of age.
2. Capable of providing informed consent and complying with study procedures.

Exclusion Criteria:

1. Any CNS diseases or psychiatric disorders (e.g., epilepsy, schizophrenia) that would interfere with study results.
2. Previous head injury.
3. Present or past (within past 6 months) drug or alcohol abuse or addiction based on DSM-5.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Motion Discrimination Performance | Study visit 1 to 2 (within a week), and study visit 3 to 4 (within a week)
  Change in accuracy on a computerized motion direction discrimination task programmed in the lab. The task assesses participants' ability to discriminate the direction of the peripherally presented moving dots at two locations (one within the blind field and the other at a mirror-symmetric location in the intact visual field). Accuracy is defined as the proportion of correct responses out of the total number of trials completed.

SECONDARY OUTCOMES:
Visual Field Change | Baseline (pre-intervention) to post-intervention follow-up (approximately 3 months, up to 6 months)
  Change in visual field function, assessed by perimetric mean deviation (PMD) measured using Humphrey perimetry. PMD is a global index representing the average deviation of visual field sensitivity compared to age-matched norms, measured in decibels (dB). More negative PMD values indicate greater visual field loss.
Visual Perception Change | Baseline (pre-intervention) to post-intervention follow-up (approximately 3 months, up to 6 months)
  Change in visual perception in the following two task:
  1. Face/Object Recognition: identify whether a peripherally presented stimulus is a face or an object.
  2. Motion Discrimination: discriminate the direction of the peripherally presented moving dots.
  Performance on both tasks will be measured at visual field locations targeted by brain stimulation and at control visual field locations not targeted by brain stimulation.
Quality of Life Change | Baseline (pre-intervention) to post-intervention follow-up (approximately 3 months, up to 6 months)
  Change in quality of life evaluated using the National Eye Institute 25 Item Visual Function Questionnaire (NEI-VFQ 25). Scores range from 0 to 100, with higher scores indicating better vision-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided